CLINICAL TRIAL: NCT05162950
Title: Effects and Importance of Epinephrine/Adrenalin Deficiency in CAH
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Anna Jung Nordenstrom, Adj Professor, Senior Consultant, Region Stockholm
Other Study IDs: CAH and epinephrine
Record Dates: First submitted 2021-12-05; First posted 2021-12-20 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood tests
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- SW CAH: Patients with 21-hydroxylase deficiency, salt wasting form.
  Interventions: Diagnostic Test: physical exercise as a standardized high intensity exercise test; Behavioral: Stress vulnerability
- SV CAH: Patients with 21-hydroxylase deficiency, simple virilising form.
  Interventions: Diagnostic Test: physical exercise as a standardized high intensity exercise test; Behavioral: Stress vulnerability
- NC CAH: Patients with 21-hydroxylase deficiency, non-classic form.
  Interventions: Diagnostic Test: physical exercise as a standardized high intensity exercise test; Behavioral: Stress vulnerability
- Carrier CAH: Healthy individuals, heterozygous carriers a mutation in the CYP21A2 gene. Recruited among parents of patients with CAH.
  Interventions: Diagnostic Test: physical exercise as a standardized high intensity exercise test; Behavioral: Stress vulnerability
- Control: Healthy sex and age matched controls
  Interventions: Diagnostic Test: physical exercise as a standardized high intensity exercise test; Behavioral: Stress vulnerability

INTERVENTIONS:
Diagnostic Test: physical exercise as a standardized high intensity exercise test — High intensity exercise test, cycling, performed at the Karolinska University Hospital
Behavioral: Stress vulnerability — Web based survey of validated psychological questionnaires measuring fatigue (MFS), exhaustion disorder (KEDS), anxiety (LSAS-SR, HADS), depression (HADS), and Karolinska sleep questionnaire
  Other Names: Validated questionnaires

SUMMARY:
Individuals with CAH produce lower levels of epinephrine (adrenalin) than controls. This can be correlated to the CYP21A2 genotype and is most pronounced in the classic forms. Individuals with CAH have an increased risk of developing hypoglycemia because both cortisol and epinephrine are important counter regulatory hormones. Stress dosing is essential in situations of increased physical stress such as infections with fever for example.

Glucocorticoid treatment and stress dosing cannot compensate fully during physical stress neither for the reaction to psychological stress. This may render various types of difficulties in the individual's life.

We aim to investigate if the deficient epinephrine production can be confirmed and if it is related to the increased level of anxiety and vulnerability to stress that we observe in the patients.

Specific aims of the study:

* Analyse the epinephrine/adrenalin production in patients with CAH using measurements of epinephrine and metanephrine in blood, during an exercise test
* Assess stress vulnerability and anxiety using validated questionnaires
* Correlate the results to severity of disease, CYP21A2 genotype
* Investigate if psychological and somatic stress symptoms are related to the epinephrine production capacity.

DETAILED DESCRIPTION:
After written informed consent study subjects, patients and controls, are invited to fill in a web based survey with the validated questionnaires. A link to the survey, expected to take 30 - 60 minutes to complete, is mailed to to the subjects . A subgroup of study subjects are invited to perform an ergo-spirometri test followed by the exercise test at the hospital. They are asked not to eat for 6 hours or drink any coffe during the day before the test. A venous catheter is used for blood sampling during the exercise. ECG, an orthostatic blood pressure test and a the ergo-spirometry test are performed before the subject is asked to do the exercise test, a cycling maximum test. Blood glucose, lactate, are followed every 4 minutes. Adrenal androgens, cortisol, insulin and methoxy-catecholamine are measured before and when the subject has reached maximum effort load and the test is ended.

The physical capacity, orthostatic blood pressure and the blood test results are related to the severity of CAH and to the maximum level of methoxy-cathecholamine produced by each individual. In the larger group of individuals, not taking part in the exercise test but completing the survey the genotype is correlated to the questionnaire results.

ELIGIBILITY:
Inclusion Criteria:

* CAH due to 21-hydroxylase deficiency,

Exclusion Criteria:

* Cardiovascular disease

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Men and women with congenital adrenal hyperplasia due to 21-hydroxylase deficienc. Sex and age matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
epinephrine level | 2022 December 31
  Measured methoxy-catecholamine at maximum exercise test, cycling test.

SECONDARY OUTCOMES:
Hospital Anxiety Depression Scale | 2022 December 31
  stress vulnerability
Mental Fatigue scale | 2022 December 31
  stress vulnerability
Liebowitz anxiety scale | 2022 December 31
  stress vulnerability
Karolinska Exhaustion disorder scale | 2022 December 31
  stress vulnerability
sleep questionnaire | 2022 December 31
  stress vulnerability

OTHER OUTCOMES:
Orthostatic blood pressure | 2022 December 31
  Blood pressure measured lying down and standing for 10 minutes
CYP21A2 genotype | 2022 December 31
  mutation analysis

CONTACTS AND LOCATIONS:
Overall Officials: Fredrika Gauffin, MDPhD, Study Director — Karolinska University Hospital
Locations (1):
- Karolinska University hospital, Stockholm, (State), Sweden